CLINICAL TRIAL: NCT03946033
Title: A Prospective Study Assessing Whether Immunoscore Colon Test Impacts the Choice of Adjuvant Chemotherapy, in a Multidisciplinary Meeting, for Treating Non-metastatic Colon Cancer Patients After Curative-intent Surgery
Brief Title: Impact of Immunoscore Colon Test on Adjuvant Therapeutic Strategy in Non-Metastatic Colon Cancer
Acronym: PROSCORE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Canceled by Immunoscore's manufacturer
Sponsor: UNICANCER (Other)
Collaborators: HalioDx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UC-0110/1813; 2018-A03339-46 (Other: ANSM)
Record Dates: First submitted 2019-05-07; First posted 2019-05-10 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Colonic Neoplasms
Keywords: Immunoscore Adjuvant Prospective Colon
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Masking Description: Immunoscore Colon Test Result will be disclosed in Multidisciplinary Meeting only after the first therapeutic decision
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): All participants are included in the same arm. Immunoscore Colon Test is applied on a tumor sample and the result is kept secret. In the Multidisciplinary Meeting evaluating the adjuvant therapy of the participant, a first therapeutic decision is taken, then Immunoscore result will be disclosed and the Multidisciplinary Meeting will take a second decision.
  Interventions: Diagnostic Test: Immunoscore Colon Test

INTERVENTIONS:
Diagnostic Test: Immunoscore Colon Test — Immunoscore Colon is a CE-marked in-vitro diagnostic test, allowing the quantification of CD3 and CD8 positive cells in formalin-fixed paraffin-embedded (FFPE) tissue samples of primary colon cancer. The test uses immunohistochemistry, digital pathology techniques and a dedicated software.

SUMMARY:
Immunoscore Colon Test (ICT) will be applied on tumor samples from curative surgery. In the Multidisciplinary Meeting (MM) evaluating the participant adjuvant strategy, a first decision will be taken, based on the participant medical record only. ICT will then be disclosed and the MM will take a second decision. The aim of the study is to observe if the ICT result modifies the treatment decision.

DETAILED DESCRIPTION:
On previous studies, Immunoscore Colon test identified subgroups of stage II and III colon cancer patients whose Chemotherapy could be adjusted.

The study hypothesis is that Immunoscore Colon Test will modify the therapeutic decision in MM.

With Alpha and Beta at 5% and p0=10% modification rate, the participating investigators need to include 280 participants, 140 in each cohort (stage II and stage III).

Participants will have tumor samples from their curative surgery tested with Immunoscore Colon. When the patients are evaluated in MM, a first therapeutic decision will be taken before disclosing the test result. ICT result will then be communicated and a second decision will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically/histologically proven colon adenocarcinoma
* non-metastatic cancer
* Stage II or III adenocarcinoma
* Surgical resection of primitive tumor within 6 weeks of multidisciplinary meeting
* No macroscopic or microscopic proof of residual disease during surgery (R0 margins)
* Available surgical material: FFPE tumor samples
* Post-operative adjuvant chemotherapy considered during multidisciplinary meeting
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Patient having signed a written informed consent prior to any trial specific procedures
* Patient affiliated to the social security system or equivalent

Exclusion Criteria:

* Other invasive cancer within 5 years of the colon cancer diagnosis, except for adequately treated basal cell carcinoma or squamous cell skin carcinoma or in sity cervical carcinoma
* Patients for which adjuvant chemotherapy is contra-indicated
* Any previous systemic or loco regional anticancer therapy for the studied colon cancer (e.g. neoadjuvant therapy)
* Patient enrolled or planned to be enrolled in another clinical trial that may influence the therapeutic decision
* Any psychological, social or geographical issue that may hinder the patient's understanding of the study or the study conduct
* Person deprived of liberty or under the authority of a legal guardian
* Person unable to understand the study or to comply with the protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Modification rate of adjuvant therapeutic strategy | At the multidisciplinary meeting, up to 6 weeks after the cancer surgery
  Modifications of adjuvant therapy, type and/or duration

CONTACTS AND LOCATIONS:
Overall Officials: David Malka, Dr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (21):
- France (21):
  - Hôpital Simone Veil, Blois
  - Hospices civils de Colmar, Colmar
  - CHU de Dijon, Dijon
  - CHD de Vendée, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Hôpital Jean Mermoz, Lyon
  - Hôpital Européen Marseille, Marseille
  - Institut Régional du Cancer de Montpellier, Montpellier
  - CHU Hôtel-Dieu, Nantes
  - Hôpital Saint-Louis, Paris
  - CHU de Bordeaux - Haut Lévêque, Pessac
  - CHU de Poitiers, Poitiers
  - Centre Hospitalier Annecy Genevois, Pringy
  - CHU de Reims, Reims
  - Centre Eugène Marquis, Rennes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Hôpital du Léman, Thonon-les-Bains
  - Institut Gustave Roussy, Villejuif
  - Hôpital privé de Villeneuve d'Ascq, Villeneuve-d'Ascq

REFERENCES:
- [Background] Pages F, Mlecnik B, Marliot F, Bindea G, Ou FS, Bifulco C, Lugli A, Zlobec I, Rau TT, Berger MD, Nagtegaal ID, Vink-Borger E, Hartmann A, Geppert C, Kolwelter J, Merkel S, Grutzmann R, Van den Eynde M, Jouret-Mourin A, Kartheuser A, Leonard D, Remue C, Wang JY, Bavi P, Roehrl MHA, Ohashi PS, Nguyen LT, Han S, MacGregor HL, Hafezi-Bakhtiari S, Wouters BG, Masucci GV, Andersson EK, Zavadova E, Vocka M, Spacek J, Petruzelka L, Konopasek B, Dundr P, Skalova H, Nemejcova K, Botti G, Tatangelo F, Delrio P, Ciliberto G, Maio M, Laghi L, Grizzi F, Fredriksen T, Buttard B, Angelova M, Vasaturo A, Maby P, Church SE, Angell HK, Lafontaine L, Bruni D, El Sissy C, Haicheur N, Kirilovsky A, Berger A, Lagorce C, Meyers JP, Paustian C, Feng Z, Ballesteros-Merino C, Dijkstra J, van de Water C, van Lent-van Vliet S, Knijn N, Musina AM, Scripcariu DV, Popivanova B, Xu M, Fujita T, Hazama S, Suzuki N, Nagano H, Okuno K, Torigoe T, Sato N, Furuhata T, Takemasa I, Itoh K, Patel PS, Vora HH, Shah B, Patel JB, Rajvik KN, Pandya SJ, Shukla SN, Wang Y, Zhang G, Kawakami Y, Marincola FM, Ascierto PA, Sargent DJ, Fox BA, Galon J. International validation of the consensus Immunoscore for the classification of colon cancer: a prognostic and accuracy study. Lancet. 2018 May 26;391(10135):2128-2139. doi: 10.1016/S0140-6736(18)30789-X. Epub 2018 May 10. PMID 29754777